CLINICAL TRIAL: NCT00250835
Title: A Phase II Trial Using a Combination of Oxaliplatin, Capecitabine, and Celecoxib With Concurrent Radiation for Patients With Newly Diagnosed Resectable Rectal Cancer
Brief Title: Combination of Oxaliplatin, Capecitabine, and Celecoxib With Concurrent Radiation for Rectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3304C; NCI-2011-02685 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2005-11-04; First posted 2005-11-08 (Estimated); Results first posted 2015-09-01 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Rectal Cancer
Keywords: Resectable Rectal Cancer; Radiation; Neoadjuvant; Rectum; GI - Colorectal Neoadjuvant; Cancer
MeSH Terms: conditions — Rectal Neoplasms; Neoplasms | interventions — Drug Therapy; Celecoxib; Radiation; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy, Celecoxib, and Radiation (Experimental): Oxaliplatin weekly at 50 mg/m2 given intravenously over two hours for the duration of radiation.
  Capecitabine: on the days of radiation at 850 mg/m2 orally twice a day [1700 mg/m2/day] (Monday through Friday during radiation therapy).
  Celecoxib at 200 mg orally twice a day throughout the duration of radiation without a break.
  Interventions: Other: Chemotherapy, Celecoxib, and Radiation

INTERVENTIONS:
Other: Chemotherapy, Celecoxib, and Radiation — Enrolled rectal cancer patients are treated with concurrent chemoradiation and celecoxib pre-operatively for at least 14 days. Definitive surgery is performed within 6 weeks from the end of treatment.
  Other Names: Celecoxib = Celebrex; Oxaliplatin = Eloxatin; Capecitabine = Xeloda

SUMMARY:
A combination of chemotherapy and radiation is often used to treat rectal cancer patients before surgery in an effort to shrink the tumor and make it easier to remove as well as to help increase the chances of sphincter-sparing surgery. Many previous clinical studies have suggested that rectal cancer patients may survive longer if the surgery results in a pathological complete response - that is, the absence of any tumor cells in the surgical specimen. However, there is still controversy over this. This study attempts to start to answer this question by treating rectal cancer patients with a combination of chemotherapy drugs (oxaliplatin and capecitabine), a cyclooxygenase-2 (COX-2) enzyme inhibitor and radiation before surgery. The rates of pathologic complete response, sphincter-sparing surgery, and disease-free survival are some of the therapeutic endpoints that will be studied.

DETAILED DESCRIPTION:
Improved regional control as demonstrated by a lower incidence of local recurrence after concurrent chemoradiation delivered either pre-operatively or post-operatively for resectable rectal cancer is supported by clinical trial data but the impact on overall survival with either approach remains controversial. An ideal regimen for preoperative chemoradiation in locally advanced rectal cancer would include agents that are both potent radio-sensitizers and effective in treating micro-metastatic disease without excessive toxicity. The cyclooxygenase-2 (COX-2) enzyme is over expressed in colorectal cancer, but the exact role of this over expression in tumorigenesis remains an active area of research. The area with the most potential in using cyclooxygenase-2 inhibitors in cancer treatment may be to use them as an adjunct to other modalities of treatment.

Taking into consideration all the above, a previous pilot trial of neoadjuvant therapy with combined oxaliplatin, capecitabine, celecoxib (a COX-2 inhibitor), and radiation was conducted in four patients with operable rectal cancer. Promising results, including pain relief and downstaging of cancer, were observed.

Therefore, this single-arm phase II trial of preoperative concurrent chemoradiation for patients with T3-4N0-2M0 rectal cancer was initiated to assess patient outcomes and explore the relationship between COX-2 expression in surgical specimens and therapeutic endpoints.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years of age or older, with biopsy proven T3-4N0-2M0 rectal cancer are eligible.
* Life expectancy of at least 2 years.
* Zubrod performance status of 0-2.
* Patients must be able to sign an informed consent.
* Adequate bone marrow function: peripheral granulocyte count of > 1,500 cells/mm3 and platelet count >100,000/mm3, hemoglobin > 10 gm/dl and absence of a regular red blood cell transfusion requirement.
* Adequate hepatic function with a total serum bilirubin < 1.5 x ULN; alkaline phosphatase, alanine aminotransferase (ALAT), and aspartate aminotransferase (ASAT) < 2.5 x the upper limit of normal (ULN); and adequate renal function as defined by a calculated creatinine clearance > 50 ml/min [Cockroft-Gault].
* Other initial cancer diagnosis more than five years ago without evidence of residual or recurrent disease
* Prior diagnosis of squamous or basal cell carcinoma of skin,no active disease at the time of enrollment.

Exclusion Criteria:

* Known metastases
* Pregnant or lactating women. Women/men of childbearing potential not using a reliable and appropriate contraceptive method.
* May receive no other concurrent chemotherapy or radiation therapy during this trial.
* Severe medical problems such as uncontrolled diabetes mellitus or cardiovascular disease or active infections
* Prior pelvic radiation
* Known active inflammatory bowel disease, Crohn's disease or ulcerative colitis.
* Medical conditions that would preclude the patient from definitive surgery at the end of concurrent chemoradiation
* Serious, uncontrolled, concurrent infection(s).
* Prior severe reaction to fluoropyrimidine therapy, or known hyper-sensitivity to 5-fluorouracil or known dihydropyrimidine dehydrogenase (DPD) deficiency.
* Treatment for other carcinomas within the last five years, except cured non-melanoma skin and treated in-situ cervical cancer.
* Participation in any investigational drug study within 4 weeks preceding the start of study treatment.
* Clinically significant cardiac disease or myocardial infarction within the last 12 months.
* History of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance of oral drug intake.
* Other serious uncontrolled medical conditions that the investigator feels might compromise study participation.
* Major surgery <4 weeks of the start of study treatment, without complete recovery.
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome.
* Known, existing uncontrolled coagulopathy
* Any of the following laboratory values:

  * Abnormal hematologic values (neutrophils < 1.5 x 10^9/L, platelet count < 100 x 10^9/L, hemoglobin < 10 gm/dl)
  * Impaired renal function (estimated creatinine clearance <50 ml/min as calculated with Cockroft-Gault equation.
  * Serum total bilirubin > 1.5 x upper normal limit.
  * ALAT, ASAT > 2.5 x upper normal limit (or > 5 x upper normal limit in the case of liver metastases).
  * Alkaline phosphatase > 2.5 x upper normal limit (or > 5 x upper normal limit in the case of liver metastases or > 10 x upper normal limit in the case of bone disease).
* Unwillingness to give written informed consent.
* Unwillingness to participate or inability to comply with the protocol for the duration of the study.
* History of allergic reactions, hypersensitivity reactions to aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs), or sulfonamides

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2005-04; Primary Completion 2012-12 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fa-Chyi Lee, MD, Principal Investigator — University of New Mexico
Locations (3):
- United States (3):
  - Hematology Oncology Associates, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico

REFERENCES:
- [Result] Araujo-Mino EP, Patt YZ, Murray-Krezan C, Hanson JA, Bansal P, Liem BJ, Rajput A, Fekrazad MH, Heywood G, Lee FC. Phase II Trial Using a Combination of Oxaliplatin, Capecitabine, and Celecoxib with Concurrent Radiation for Newly Diagnosed Resectable Rectal Cancer. Oncologist. 2018 Jan;23(1):2-e5. doi: 10.1634/theoncologist.2017-0474. Epub 2017 Nov 20. PMID 29158365
- See also: University of New Mexico Cancer Center — http://www.cancer.unm.edu
- See also: New Mexico Cancer Care Alliance — http://www.nmcca.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from participating cancer clinics across the state of New Mexico
Groups:
- Chemotherapy, Celecoxib, and Radiation: Oxaliplatin weekly at 50 mg/m2 given intravenously over two hours for the duration of radiation.
  Capecitabine: on the days of radiation at 850 mg/m2 orally twice a day [1700 mg/m2/day] (Monday through Friday during radiation therapy).
  Celecoxib at 200 mg orally twice a day throughout the duration of radiation without a break.
  Chemotherapy, Celecoxib, and Radiation: Enrolled rectal cancer patients are treated with concurrent chemoradiation and celecoxib pre-operatively for at least 14 days. Definitive surgery is performed within 6 weeks from the end of treatment.
Period: Overall Study
Arm/Group | Chemotherapy, Celecoxib, and Radiation
Started | 38
Completed | 37
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Chemotherapy, Celecoxib, and Radiation
Number analyzed (Participants) | 37
Age, Continuous [Mean (Full Range); unit: years] | 52 [20 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response (PCR)
Description: The pathologic complete response (PCR) rate will be calculated as the proportion of patients who achieve complete response out of all evaluable patients. PCR is defined as the total absence of residual tumor cells by microscopic examination of the resected surgical specimen, including all of the sampled lymph nodes.
Time Frame: At surgery (up to 6 weeks after end of treatment)
Population: Patients who continue on at least two of the three drugs for a minimum of 14 days are considered evaluable for the primary objective
Measure: Number (95% Confidence Interval); unit: percentage of evaluable participants
Arm/Group | Chemotherapy, Celecoxib, and Radiation
Number analyzed (Participants) | 32
percentage of evaluable participants | 31 [16 to 50]

2. Secondary Outcome: Toxicity
Description: All toxicities encountered during the study will be evaluated according to the grading system (0-5) NCI CTCAE (Common Terminology Criteria for Adverse Events) version 3.0.
  Toxicity will be reported as the proportion of subjects experiencing Grades 3,4, and 5 adverse events (AEs) out of all evaluable patients
Time Frame: Up to 3 years
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy, Celecoxib, and Radiation
Number analyzed (Participants) | 32
percentage of participants
  Grade 3 and 4 diarrhea | 9
  Grade 3 and 4 abnormal liver function tests | 9
  Grade 3 and 4 abdominal pain | 6
  Death (from severe infection) | 6

3. Secondary Outcome: Progression-free Survival (PFS)
Description: The Response Evaluation Criteria In Solid Tumors (RECIST) guidelines (Version 1.0) will be used to determine tumor response and progression. Progressive disease (PD) for target lesions: >= 20% increase in the sum of diameters of the target lesions taking as reference the smallest sum on study, and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered . PD for non-target lesions is defined as unequivocal appearance of one or more new malignant lesions or unequivocal progression of existing non-target lesions. Time to progression will be measured from the time of surgery or clinically documented down staging if surgery for whatever reason is not carried in the subject until there is evidence of PD.
  Progression-free survival is reported as the percentage of patients who have not experienced progression of disease at three years post-surgery
Time Frame: 3 years after surgery
Measure: Number (95% Confidence Interval); unit: percentage of evaluable participants
Arm/Group | Chemotherapy, Celecoxib, and Radiation
Number analyzed (Participants) | 32
percentage of evaluable participants | 84 [65 to 93]

4. Secondary Outcome: Incidence of Sphincter-sparing Surgery
Description: Incidence of sphincter-saving surgery is defined as the proportion of subjects who do not have permanent colostomy at the final follow-up out of all evaluable patients.
Time Frame: At surgery (up to 6 weeks after end of treatment)
Measure: Number (95% Confidence Interval); unit: percentage of evaluable participants
Arm/Group | Chemotherapy, Celecoxib, and Radiation
Number analyzed (Participants) | 32
percentage of evaluable participants | 56 [38 to 74]

5. Secondary Outcome: Surgical Downstaging Rate
Description: Downstaging rate after neoadjuvant treatment with combination oxaliplatin, capecitabine, celecoxib and concurrent radiation is defined as the proportion of patients whose pathological stage (stage at surgery) is different from their clinical stage (stage at baseline)
Time Frame: At surgery (up to 6 weeks after treatment)
Measure: Number (95% Confidence Interval); unit: percentage of evaluable participants
Arm/Group | Chemotherapy, Celecoxib, and Radiation
Number analyzed (Participants) | 32
percentage of evaluable participants | 75 [57 to 89]

6. Secondary Outcome: Pelvic Local Control Rate
Description: Pelvic local control rate is defined as the proportion of subjects who have no evidence of pelvic recurrence (by standard clinical assessment, including CT scan and clinical examination) at the final follow-up evaluation, out of all evaluable patients
Time Frame: Up to 3 years after surgery
Measure: Number; unit: percentage of evaluable participants
Arm/Group | Chemotherapy, Celecoxib, and Radiation
Number analyzed (Participants) | 32
percentage of evaluable participants | 6

ADVERSE EVENTS:
Arm/Group | Chemotherapy, Celecoxib, and Radiation
Serious Adverse Events (participants affected / at risk) | 6/37
Other Adverse Events (participants affected / at risk) | 29/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy, Celecoxib, and Radiation (N=37)
Dehydration (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Opportunistic Infection (Infections and infestations) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy, Celecoxib, and Radiation (N=37)
Hemoglobin decreased (Blood and lymphatic system disorders) | 5 (5)
Leukocytes decreased (Blood and lymphatic system disorders) | 3 (12)
Lymphocytes decreased (Blood and lymphatic system disorders) | 4 (15)
Platelets decreased (Blood and lymphatic system disorders) | 2 (4)
Fatigue (General disorders) | 13 (18)
Weight loss (General disorders) | 5 (7)
Decubitus ulcer (skin breakdown) (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis due to radiation (Skin and subcutaneous tissue disorders) | 6 (6)
Pruritus (Itching) (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Anorexia (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 5 (5)
Dehydration (Gastrointestinal disorders) | 5 (6)
Diarrhea (Gastrointestinal disorders) | 18 (27)
Nausea (Gastrointestinal disorders) | 14 (22)
Vomiting (Gastrointestinal disorders) | 3 (5)
Rectal hemorrhage (Gastrointestinal disorders) | 3 (4)
Hyperbilirubinemia (Investigations) | 2 (7)
Hyperglycemia (Investigations) | 2 (4)
Hypoalbuminemia (Investigations) | 7 (12)
Hypocalcemia (Investigations) | 4 (9)
Hypokalemia (Investigations) | 5 (7)
Hypomagnesemia (Investigations) | 3 (3)
Hyponatremia (Investigations) | 3 (3)
Increased blood urea nitrogen (Investigations) | 2 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 4 (4)
Insomnia (Nervous system disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 9 (12)
Abdominal pain (General disorders) | 8 (8)
Pain (General disorders) | 2 (2)
Pain in extremity (General disorders) | 3 (3)
Rectal pain (General disorders) | 6 (7)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cystitis (bladder inflammation) (Renal and urinary disorders) | 2 (2)
Dysuria (painful urination) (Renal and urinary disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes